CLINICAL TRIAL: NCT06681519
Title: The Effectiveness of Acupressure on the Physiological and Psychological Improvement of Patients Undergoing Local Anesthesia
Acronym: LA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yu-Jui Feng (Other)
Responsible Party: Sponsor-Investigator, Yu-Jui Feng, postgraduate, National Taipei University of Nursing and Health Sciences
Organization: National Taipei University of Nursing and Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Local Anesthesia; MMH IRB (Other: MMH)
Record Dates: First submitted 2024-09-16; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Assessing the Effect of Acupoint Massage on Pain and Anxiety in Patients Undergoing Surgery Under Local Anesthesia
Keywords: Key words: local anaesthesia , acupressure, physiology, psychology, autonomic nerve system

STUDY DESIGN:
Intervention Model Description: Research model type: Indicate whether parallel group design, crossover design, causal comparison, etc. are used. For example: "This study uses a parallel group design, randomly assigning subjects to the experimental group and the control group."
  Details of the intervention model: If different intervention approaches or multiple intervention groups are involved, you can describe the details of each intervention group. For example: "The experimental group received specific acupoint massage (Hegu LI4, Shenmen HT7), and the control group received standard care."
  Allocation and randomization methods: Describe the allocation method, such as random assignment or stratified randomization.
  Experimental controls: If there are control groups, placebo controls, or other controls, you can state this here.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): Acupoint pressure Group 1relieves pain and anxiety pain .
  Interventions: Procedure: Experimental Group 1 - Acupoint Pressure Experimental Group 2 - Pressure Ball Control Group - Conventional Treatment
- Group 2 (Active Comparator): Holding a pressure ball Group 2reduces pain and anxiety pain.
  Interventions: Procedure: Experimental Group 1 - Acupoint Pressure Experimental Group 2 - Pressure Ball Control Group - Conventional Treatment
- Group 3 (Sham Comparator): conventional group 3 treatmente.
  Interventions: Procedure: Experimental Group 1 - Acupoint Pressure Experimental Group 2 - Pressure Ball Control Group - Conventional Treatment

INTERVENTIONS:
Procedure: Experimental Group 1 - Acupoint Pressure Experimental Group 2 - Pressure Ball Control Group - Conventional Treatment — Interventions Group 1 - Acupoint Pressure Group 2 - Hand-Held Pressure Ball Control Group 3 - Conventional Treatment Other Names: Stress ball holding, acupoint pressure, conventional treatment
  Description: Before the intervention, subjects completed a pre-test. Afterward, they assumed a relaxed, comfortable lying position. The examiner applied acupoint pressure at four specific points: Hegu (LI4), Shenmen (HT7), Neiguan (PC6), and Zhongchong (PC9).
  The technique involves using the thumb pad to apply circular and vertical pressure on each acupoint, with the other four fingers stabilizing against the skin to ensure even pressure. The pressure is gradually increased from light to moderate until the patient experiences sensations of soreness, numbness, or swelling, commonly described as deqi (Ye Meiling et al., 2020).
  Each acupoint is pressed vertically for 3 seconds, then rotated clockwise at a rate of 2-3 rotations per second for another 3 second
  Other Names: Experimental Group 1 - Acupoint Pressure： Other Names: 「穴位按壓」、「Acupressure」 Experimental Group 2 - Pressure Ball： Other Names: 「Holding stress ball in hand」、「握壓力球」、「壓力球療法」 Control Group - Convention

SUMMARY:
Background: Local anaesthesia surgeries are outpatient procedures that allow patients to go home the same day. However, these surgeries often cause pain and anxiety for patients. Opioids are commonly used for pain management, but concerns about allergies and side effects have driven the need for alternative, safer treatments. Traditional Chinese medicine emphasizes the meridian system, which regulates qi, energy, and blood flow in the body. Stimulating acupoints on these meridians may help alleviate various ailments. This study examines whether acupressure can reduce pain and anxiety and improve physiological outcomes in patients undergoing local anaesthesia.

Objective: To assess the effectiveness of acupressure on reducing pain and anxiety, and enhancing physiological outcomes in local anaesthesia patients.

Methods: A randomized controlled trial was conducted with adult patients under local anaesthesia. The experimental group received acupressure at specific points (Hegu LI4 and Shenmen HT7), while the control group received standard care. Pain, anxiety, and autonomic function were measured before and after the intervention using IBMSPSS version 20.0 for analysis.

DETAILED DESCRIPTION:
Summary:

Outpatient surgeries with local anesthesia allow patients to return home the same day but can often lead to pain and anxiety. Although opioids are frequently used for pain management, concerns about allergies and side effects prompt the search for safer alternatives. Traditional Chinese medicine (TCM) suggests that stimulating acupoints along the body's meridian system can promote the flow of qi, energy, and blood, potentially alleviating various ailments. This study investigates whether acupressure can effectively reduce pain, anxiety, and improve physiological outcomes in patients undergoing local anesthesia.

Objective: To determine if acupressure can reduce pain and anxiety while improving physiological outcomes in patients receiving local anesthesia.

Methods: A randomized controlled trial was conducted with adults undergoing local anesthesia. The experimental group received acupressure on the Hegu (LI4) and Shenmen (HT7) points, while the control group received standard care. Pain, anxiety, and autonomic function were measured before and after the intervention, analyzed using IBM SPSS version 20.0.

Additional Context: Distraction techniques, including VR, music, videos, breathing exercises, vibration stimulation, and acupressure with hand-held pressure balls, have been shown to help patients manage pain and anxiety during procedures. This study uses acupressure and pressure balls to create a positive psychological model for managing stress, fear, and anxiety, potentially helping patients adopt a better mental approach toward surgery.

ELIGIBILITY:
1. The acceptance conditions of the subject must meet:

1. Adults (20-64 years old).
2. Mainly patients receiving local anesthesia.
3. Those who have no abnormal limb sensation and good skin integrity, and can perform normal acupoint pressure.
4. Those who are willing to participate in this study and can communicate in Mandarin and Taiwanese.

2. Exclusion conditions:

1. Those who have taken painkillers before surgery.
2. The surgical site is already inflamed.
3. Those diagnosed with mental illness and cognitive impairment.
4. Heart disease and arrhythmia (pacemaker).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
The Effectiveness of Acupressure on the Physiological and Psychological Improvement of Patients Undergoing Local Anesthesia | This study used Visual Analogue Scales (VAS) to measure patient pain. Divide a straight line about 10 centimeters into 10 equal parts from left to right. The left side is 0 points, no pain at all, and the right side is 10 points, very painful. Ask the su
  Acupressure relieves pain and relieves anxiety
The Effectiveness of Acupressure on the Physiological and Psychological Improvement of Patients Undergoing Local Anesthesia | Heart rate variability (HRV, Heart Rate Variability) in patients undergoing local anesthesia surgery refers to the change in heartbeat intervals. High HRV is generally considered a sign of health, meaning that the heart is able to flexibly respond to var
  Acupressure with HRV
The Effectiveness of Acupressure on the Physiological and Psychological Improvement of Patients Undergoing Local Anesthesia | This study used the Chinese version of The State-Trait Anxiety Inventory (STAI-6) to measure the patient's anxiety state. The Short State-Trait Anxiety Inventory-6 (Short State-Trait Anxiety Inventory-6) consists of 6 questions selected from the STAI on
  Physiological effects

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Yu Jui Feng, Taipei, Taiwan
  - YuJui Feng, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
This study needs to be reviewed by the hospital's clinical ethics committee before it can be accepted. The written informed consent form is signed and dated, and the researcher's contact information is clearly stated on the consent form. Participants can terminate participation in the study at any time. After all participants agree and sign a written consent form, they will fulfill their confidentiality responsibilities. Subject information will be replaced with personal information by codes to protect subject privacy. The case data are collected, each case is individually coded and locked in a designated cabinet. The key holder of the cabinet is the researcher. After the research data are kept for two years, they are shredded with a fine shredder and discarded.

REFERENCES:
- See also: https://pubmed.ncbi.nlm.nih.gov/?term=%231+AND+%235&amp;amp;amp;sort=date&amp;amp;amp;filter=pubt.randomizedcontrolledtrial&amp;amp;amp;filter=pubt.randomizedcontrolledtrial — https://pubmed.ncbi.nlm.nih.gov/?term=%231+AND+%235&amp;amp;amp;sort=date&amp;amp;amp;filter=pubt.randomizedcontrolledtrial&amp;amp;amp;filter=pubt.randomizedcontrolledtrial